CLINICAL TRIAL: NCT01273038
Title: Clinical Investigation of Filter Improvement for New Filter to Ostomy Bags
Brief Title: Clinical Investigation for New Filter to Ostomy Bags
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP210OC
Record Dates: First submitted 2010-12-14; First posted 2011-01-10 (Estimated); Results first posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2012-11

CONDITIONS: Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SenSura (Active Comparator): The reference product is the CE marked and launched SenSura product which is commercially available
  Interventions: Device: SenSura
- Morfeus (Experimental): The test product is the product with the proposed new Morfeus filter
  Interventions: Device: Morfeus

INTERVENTIONS:
Device: Morfeus — The new ostomy bag filter (called Morfeus) will be tested for a period of 14 days
  Arms: Morfeus
Device: SenSura — The CE marked ostomy bag filter will be tested for a period of 14 days
  Arms: SenSura

SUMMARY:
The aim of the current clinical investigation is to evaluate a new filter.

DETAILED DESCRIPTION:
The new filter has been developed in order to significantly reduce problems with ballooning and other problems related to filter performance in people with a stoma.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and have full legal capacity.
* Have given written informed consent.
* Be able to fill in the Case Report Form.
* Be colostomy operated and have had a stoma for at least 6 months.
* Experience ballooning at least once per week.
* Be able to manage the bags themselves (application, removal).
* Be able to use a flat base plate.
* Have a stoma with a diameter less than 60 mm

Exclusion Criteria:

* Persons who irrigate
* Currently suffer from peristomal skin problems (i.e. bleeding or broken skin).
* Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
* Pregnant or breastfeeding.
* Participate in other test at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, MSc, Study Chair — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a user database in Denmark
Pre-assignment Details: 20 subjects were enrolled and randomized in the study
Groups:
- Morfeus First (Test Filter), Then SenSura (Reference Filter): First Intervention with Morfeus (14 days) then Second Intervention with SenSura (14 days)
- SenSura First (Reference Filter), Then Morfeus (Test Filter): First Intervention with SenSura (14 days) then Second Intervention with Morfeus (14 days)
Period: First Intervention (14 Days)
Arm/Group | Morfeus First (Test Filter), Then SenSura (Reference Filter) | SenSura First (Reference Filter), Then Morfeus (Test Filter)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Morfeus First (Test Filter), Then SenSura (Reference Filter) | SenSura First (Reference Filter), Then Morfeus (Test Filter)
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Morfeus (Test Filter): The new filter Morfeus is intended to clean the air and prevent ballooning in a 1-piece colostomy appliance.
- SenSura (Reference Filter): The reference filter was the commercially available Sensura filter on the 1-piece colostomy bag.
- Total: Total of all reporting groups
Arm/Group | Morfeus (Test Filter) | SenSura (Reference Filter) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 66 (7) | 66 (6)
Sex/Gender, Customized [Number; unit: participants]
  Female | 3 | 5 | 8
  Male | 6 | 5 | 11
  Gender information not available | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Ballooning in the Morfeus and SenSura Test Period.
Description: Data will not be recorded at specific time points due to individual changing patterns (1-3 bags per day). Study subjects will fill out the Case Report Form (CRF) by themselves when changing bag. The subject is asked in the CRF among others the reason for changing bag (e.g. ballooning). Subjects will change bag according to their normal routine or when deemed appropriate. They are advised to change bag if it is filled with air and the air cannot be released through the filter within a specified time period.
Time Frame: Daily or at every change of bag in a period of a maximum of 28 days
Population: ITT
Measure: Number; unit: percentage of bags
Units Other Than Participants: bags
Arm/Group | Morfeus (Test Filter) | SenSura (Reference Filter)
Number analyzed (Participants) | 20 | 20
Number analyzed (bags) | 526 | 567
percentage of bags | 23 | 11

ADVERSE EVENTS:
Arm/Group | Morfeus (Test Filter) | SenSura (Reference Filter)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morfeus (Test Filter) (N=20) | SenSura (Reference Filter) (N=20)
Skin redness and puritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes